CLINICAL TRIAL: NCT00685516
Title: Effects of Brewed Green and Black Tea on Inflammation, Apoptosis and Oxidation in Men With Prostate Cancer
Brief Title: Green Tea, Black Tea, or Water in Treating Patients With Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-001050; R01CA116242 (NIH); UCLA-061109702 (Other: UCLA); CDR0000596162 (Other: UCLA)
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I - Green Tea (Active Comparator): Patients receive 6 cups of green tea daily for 2-8 weeks in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: green tea
- Arm II - Water (Placebo Comparator): Patients receive 6 cups of water daily for 2-8 weeks in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: placebo
- Arm III - Decaffeinated black tea (Active Comparator): Patients receive 6 cups of decaffeinated black tea daily for 2-8 weeks in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: decaffeinated black tea

INTERVENTIONS:
Dietary Supplement: green tea — 6 cups of green tea daily for 2-8 weeks
  Arms: Arm I - Green Tea
Dietary Supplement: placebo — 6 cups of water daily for 2-8 weeks
  Arms: Arm II - Water
Dietary Supplement: decaffeinated black tea — 6 cups of decaffeinated black tea daily for 2-8 weeks
  Arms: Arm III - Decaffeinated black tea

SUMMARY:
RATIONALE: Green tea contains ingredients that may prevent or slow the growth of certain cancers. It is not yet known whether green tea is more effective than black tea or water in treating prostate cancer.

PURPOSE: This randomized phase II trial is studying green tea to see how well it works compared with black tea and water in treating patients with prostate cancer undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* to determine the effect of GT and BT consumption on apoptosis (TUNEL, ratio Bax:Bcl-2), proliferation, oxidation, and inflammation in malignant radical prostatectomy tissue compared to water control using immunohistochemistry.
* to examine levels of tea polyphenols and methylated tea polyphenol metabolites in fresh frozen radical prostatectomy tissue and urine, urinary oxidative DNA damage (8OHdG) and serum prostate-specific antigen (PSA) levels.

OUTLINE: This is a multicenter, randomized study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive 6 cups of green tea daily for 2-8 weeks in the absence of unacceptable toxicity.
* Arm II: Patients receive 6 cups of water daily for 2-8 weeks in the absence of unacceptable toxicity.
* Arm III: Patients receive 6 cups of decaffeinated black tea daily for 2-8 weeks in the absence of unacceptable toxicity.

Patients undergo radical prostatectomy.

Blood and urine samples, as well as tissue from diagnostic biopsy and radical prostatectomy specimens, are obtained for laboratory correlative studies. Samples are assessed by IHC, high-performance liquid chromatography, or mass spectrometry for changes in prostate tumor grade, stage, and margin status; concentrations of total and free tea polyphenols (i.e., EGCG, EC, EGC, ECG), theaflavins, and conjugated/colonic tea metabolites; biomarkers of prostate cancer development and progression (i.e., serum PSA, proliferation [i.e., Ki-67], apoptosis [i.e., TUNEL, Bax/Bcl-2 ratio], inflammation [i.e., NFkB]), and oxidative status (i.e., 8OhdG/dG ratio); and genotype and gene expression of metabolizing enzymes (i.e., COMT, UGT, and SULT). Serum samples are also assessed by ex vivo LNCaP cell culture assay for antiproliferative activity and by competitive chemiluminescent immunoassay for concentrations of PSA, IGF-1, IGFBP-3, testosterone, SHBG, and DHEA-sulfate.

ELIGIBILITY:
Inclusion Criteria:

* subject consents to participate in the trial.
* subject is 40-75 years of age and has a diagnosis of adenocarcinoma of the prostate.
* Scheduled to undergo radical prostatectomy.
* The subject agrees to stop consumption of tea or tea-containing products throughout the entire intervention period except for the tea provided during study intervention.
* The subject agrees to stop consumption of dietary or vitamin supplements (e.g., lycopene, Vitamin E, selenium, genistein) or herbal supplements (e.g., saw palmetto, PC-SPES)

Exclusion Criteria:

* history of hepatitis or liver dysfunction
* ongoing alcohol abuse
* significant medical or psychiatric conditions that would make the patient a poor protocol candidate
* prior sensitivity or allergic reaction to tea, tea products, or tea supplements
* allergy or sensitivity to multiple food items or nutritional supplements
* concurrent luteinizing hormone-releasing hormone agonists, androgen receptor blocking agents, or finasteride
* prior bilateral orchiectomy

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2012-01-12 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M. Henning, PhD, RD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California

REFERENCES:
- [Result] Henning SM, Wang P, Said JW, Huang M, Grogan T, Elashoff D, Carpenter CL, Heber D, Aronson WJ. Randomized clinical trial of brewed green and black tea in men with prostate cancer prior to prostatectomy. Prostate. 2015 Apr 1;75(5):550-9. doi: 10.1002/pros.22943. Epub 2014 Dec 24. PMID 25545744

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea
Started | 42 | 38 | 33
Completed | 34 | 33 | 26
Not Completed | 8 | 5 | 7

BASELINE CHARACTERISTICS:
Population: 93 subjects completed the intervention (Arm I, GT: 34, Arm II, control: 33, Arm III, BT: 26).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea | Total
Number analyzed (Participants) | 34 | 33 | 26 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (6.9) | 61.8 (6.2) | 61.4 (7.4) | 61.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 34 | 33 | 26 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 6 | 18
  White | 27 | 23 | 13 | 63
  More than one race | 1 | 3 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 26 | 93
Weight (KG) [Mean (Standard Deviation); unit: kg] | 85.7 (12.2) | 86.6 (14.3) | 89.9 (13.4) | 87.6 (14)
Height (cm) [Mean (Standard Deviation); unit: cm] | 176 (21) | 175 (22) | 175 (22) | 175.3 (22)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (3.8) | 27.4 (4.9) | 27.4 (3.6) | 27.3 (4)
Biopsy Gleason Score (percent) [Number; unit: participants] — Gleason Score: a system of grading prostate cancer tissue based on how it looks under a microscope. Gleason scores range from 2 to 10 and indicate how likely it is that a tumor will spread. A low Gleason score means the cancer tissue is similar to normal prostate tissue and the tumor is less likely to spread; a high Gleason score means the cancer tissue is very different from normal and the tumor is more likely to spread. A score of Gleason 7 (3 + 4) is considered significantly better and the cancer less likely to spread then a Gleason score of 7 (4 + 3).
  participants
    6 | 18 | 12 | 11 | 41
    7 (3+4) | 9 | 15 | 9 | 33
    7 (4+3) | 3 | 3 | 3 | 9
    greater than or equal to 8 | 4 | 3 | 3 | 10
Serum prostate-specific antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 9.6 (5.2) | 9.9 (8.5) | 9.2 (4.3) | 9.6 (6)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Green Tea (GT) and Black Tea (BT) Consumption on Percentage of Cells With Positive Staining for Apoptosis, Proliferation, Oxidation, and Inflammation in Malignant Radical Prostatectomy Tissue Compared to Water Control Using Immunohistochemistry.
Description: To determine the effect of Green Tea and Black Tea consumption on Prostate cancer tissue by examining programmed cell death, cell proliferation, cell oxidation, and cellular inflammation in that malignant radical prostatectomy tissue compared to water control using immunohistochemistry.
Time Frame: 6 weeks
Population: subjects that completed study
Measure: Mean (Standard Deviation); unit: percent positive of total cells
Groups:
- Arm II - Water: Placebo:patients receive 6 cups of water daily for 2-8 weeks in the absence of unacceptable toxicity.
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea
Number analyzed (Participants) | 34 | 33 | 26
percent positive of total cells
  Staining proliferation (Ki67) | 2.48 (1.83) | 2.3 (1.55) | 4.38 (4.1)
  Staining apoptosis Tunel | 6.96 (8.56) | 6.7 (9.1) | 6.57 (8.85)
  Staining oxidative DNA Damage 8OHdG | 5.5 (7.4) | 7.27 (10.68) | 11.23 (12.01)
  Staining Proliferation Bax | 37.4 (11) | 37.06 (8.71) | 37.35 (7.58)
  Staining Proliferation Bcl-2 | 2.92 (2.97) | 5.21 (6.91) | 6.48 (6.25)
  NFKB cytoplasmic staining | 21.23 (20.46) | 22.3 (14.62) | 19.21 (14.63)
  NFkB nuclear staining | 1.46 (1.79) | 5.13 (6.37) | 4.58 (6.61)

2. Secondary Outcome: Concentration of Tea Polyphenols, Their Metabolites, and Colonic Metabolites in Prostate Tissue
Description: Examine levels of tea polyphenols and methylated tea polyphenol metabolites in fresh frozen radical prostatectomy tissue and urine, urinary oxidative DNA damage (8OHdG) and serum prostate-specific antigen (PSA) levels.
Time Frame: 6 weeks
Population: Concentration of tea polyphenols and methyl-metabolites in prostate tissue after the consumption of GT and BT. No polyphenols were found after water consumption.
  (-)-epigallocatechin-3-gallate (EGCG), (-)-epicatechin-3-gallate (ECG), (-)-epigallocatechin (EGC) , (-)-epicatechin (EC), 4'-O-methylEGC (4'-MeEGC), 4"-O-methylEGCG (4"-OmethylEGCG).
Measure: Mean (Standard Deviation); unit: (pmol/g tissue)
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea
Number analyzed (Participants) | 34 | 33 | 26
(pmol/g tissue)
  EGCG | 42.1 (32.4) | 0 (0) | 0 (0)
  ECG | 17.8 (10.1) | 0 (0) | 0 (0)
  4" MeEGCG | 38.9 (19.5) | 0 (0) | 0 (0)
  Theaflavin | 0 (0) | 0 (0) | 0 (0)

3. Secondary Outcome: Concentration of Tea Polyphenols and Methyl-metabolites in Urine After the Consumption of Green Tea (GT) and Black Tea (BT).
Description: Concentration of tea polyphenols and methyl-metabolites in urine after the consumption of GT and BT. No polyphenols were found after water consumption
Time Frame: 6 weeks
Population: Urine concentration of (-)-epigallocatechin-3-gallate (EGCG), (-)-epicatechin-3-gallate (ECG), (-)-epigallocatechin (EGC) , (-)-epicatechin (EC), 4'-O-methylEGC (4'-MeEGC), 4"-O-methylEGCG (4"-OmethylEGCG).
Measure: Mean (Standard Deviation); unit: umol/g creatinine
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea
Number analyzed (Participants) | 34 | 33 | 26
umol/g creatinine
  EGC | 9.2 (16) | 0 (0) | .4 (.4)
  EC | 4.8 (6.1) | 0 (0) | .3 (.3)
  4'-MeEGC | 8.0 (18) | 0 (0) | .2 (.3)
  Theaflavins | 0 (0) | 0 (0) | 0 (0)

4. Secondary Outcome: Prostate Specific Antigen (PSA) After the Consumption of Green Tea (GT) and Black Tea (BT).
Time Frame: 6 weeks
Population: Pre and post blood samples unavailable for: 4 participants in Arm I (GT group), 3 participants in Arm II (control/water group) and 3 participants in Arm III (BT group).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea
Number analyzed (Participants) | 30 | 30 | 23
ng/mL | 8.4 (4.3) | 10.0 (9.0) | 9.6 (6.0)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Arm I - Green Tea | Arm II - Water | Arm III - Decaffeinated Black Tea
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/26
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No